CLINICAL TRIAL: NCT06670898
Title: A Phase 1, Open-label Study of the Absorption, Metabolism, Excretion of [14C]-NS-580 Following a Single Oral Dose in Healthy Male Subjects
Brief Title: A Study of Absorption, Metabolism, Excretion of [14C]-NS-580 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nippon Shinyaku Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NS580-P1-06
Record Dates: First submitted 2024-10-22; First posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Administration of [14C] NS-580 (Experimental)
  Interventions: Drug: [14C] NS-580

INTERVENTIONS:
Drug: [14C] NS-580 — Oral suspension

SUMMARY:
The purpose of this study was to determine the absorption, metabolism, and excretion of radioactivity and to characterize and determine, where possible, the metabolites present in plasma, urine, and faeces in healthy male subjects following a single oral administration of [14C]-NS-580.

ELIGIBILITY:
Inclusion Criteria:

* Males of any race, between 35 and 60 years of age, inclusive.
* Body mass index between 18.0 and 32.0 kg/m2, inclusive.
* History of a minimum of 1 bowel movement per day.

Exclusion Criteria:

* Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, haematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the investigator (or designee).
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the investigator (or designee).

Ages: 35 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2023-11-08 (Actual); Primary Completion 2024-01-18 (Actual); Study Completion 2024-01-18 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve, from time 0 infinity (AUC0-inf) of NS-580 in plasma | Pre-dose up to 28 days post-dose
  AUC0-inf of NS-580 in plasma
AUC0-inf of [14C] NS-580 in plasma and whole blood for Total Radioactivity | Pre-dose up to 56 days post-dose
  AUC0-inf of [14C] NS-580 in plasma and whole blood
Area under the concentration-time curve from time 0 to the time of the last quantifiable concentration (AUC0-tlast) | Pre-dose up to 28 days post-dose
  AUC0-tlast of NS-580 in plasma
AUC0-tlast of [14C] NS-580 in plasma and whole blood for Total Radioactivity | Pre-dose up to 56 days post-dose
  AUC0-tlast of [14C] NS-580 in plasma and whole blood
Maximum observed concentration (Cmax) of NS-580 | Pre-dose up to 28 days post-dose
  Cmax of NS-580 in plasma
Cmax of [14C] NS-580 in plasma and whole blood for Total Radioactivity | Pre-dose up to 56 days post-dose
  Cmax of [14C] NS-580 in plasma and whole blood
Time of the maximum observed concentration (Tmax) of NS-580 | Pre-dose up to 28 days post-dose
  Tmax of NS-580 in plasma
Tmax of [14C] NS-580 in plasma and whole blood for Total Radioactivity | Pre-dose up to 56 days post-dose
  Tmax of [14C] NS-580 in plasma and whole blood
Apparent terminal elimination half-life (t1/2) of NS-580 | Pre-dose up to 28 days post-dose
  t1/2 of NS-580 in plasma
t1/2 of [14C] NS-580 in plasma and whole blood for Total Radioactivity | Pre-dose up to 56 days post-dose
  t1/2 of [14C] NS-580 in plasma and whole blood
Renal clearance (CLR) of NS-580 | Pre-dose up to 28 days post-dose
  CLR of NS-580 in plasma
Amount of dose administered urine recovered (Aeu) of NS-580 | Pre-dose up to 56 days post-dose
  Aeu of NS-580
Percentage of dose administered urine recovered (feu) of NS-580 | Pre-dose up to 56 days post-dose
  feu of NS-580
Total radioactivity recovery | Pre-dose up to 56 days post-dose
  Total radioactivity recovery in urine and faeces

SECONDARY OUTCOMES:
Proportions of NS-580 major metabolites | Pre-dose up to 56 days post-dose
Incidence and severity of AEs | Pre-dose up to 56 days post-dose

CONTACTS AND LOCATIONS:
Locations (1):
- Fortrea Clinical Research Unit Ltd, Leeds, United Kingdom